CLINICAL TRIAL: NCT04145115
Title: A Phase II Study of Checkpoint Blockade Immunotherapy in Patients With Somatically Hypermutated Recurrent WHO Grade 4 Glioma
Brief Title: A Study Testing the Effect of Immunotherapy (Ipilimumab and Nivolumab) in Patients With Recurrent Glioma With Elevated Mutational Burden
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2019-07242; NCI-2019-07242 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); A071702 (Other: Alliance for Clinical Trials in Oncology); A071702 (Other: CTEP); U10CA180821 (NIH)
Record Dates: First submitted 2019-10-29; First posted 2019-10-30 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Astrocytoma, IDH-Mutant, Grade 4; Diffuse Glioma; Glioblastoma, IDH-Wildtype; Secondary Glioblastoma
MeSH Terms: conditions — Astrocytoma; Glioblastoma | interventions — Ipilimumab; CTLA-4 Antigen; Magnetic Resonance Spectroscopy; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (nivolumab, ipilimumab) (Experimental): Patients receive nivolumab IV over 30 minutes and ipilimumab IV over 30 minutes on day 1. Treatment repeats every 3 weeks for 4 cycles in the absence of disease progression or unacceptable toxicity. Patients then receive nivolumab IV over 30 minutes on day 1. Cycles repeat every 4 weeks in the absence of disease progression or unacceptable toxicity. Patients also undergo MRI throughout the study.
  Interventions: Biological: Ipilimumab; Procedure: Magnetic Resonance Imaging; Biological: Nivolumab

INTERVENTIONS:
Biological: Ipilimumab — Given IV
  Other Names: Anti-Cytotoxic T-Lymphocyte-Associated Antigen-4 Monoclonal Antibody; BMS 734016; BMS-734016; BMS734016; Ipilimumab Biosimilar CS1002; MDX 010; MDX-010; MDX-CTLA4; MDX010; Yervoy
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Biological: Nivolumab — Given IV
  Other Names: ABP 206; BCD-263; BMS 936558; BMS-936558; BMS936558; CMAB819; MDX 1106; MDX-1106; MDX1106; NIVO; Nivolumab Biosimilar ABP 206; Nivolumab Biosimilar BCD-263; Nivolumab Biosimilar CMAB819; ONO 4538; ONO-4538; ONO4538; Opdivo

SUMMARY:
This phase II trial studies the effect of immunotherapy drugs (ipilimumab and nivolumab) in treating patients with glioma that has come back (recurrent) and carries a high number of mutations (mutational burden). Cancer is caused by changes (mutations) to genes that control the way cells function. Tumors with high number of mutations may respond well to immunotherapy. Immunotherapy with monoclonal antibodies such as ipilimumab and nivolumab may help the body's immune system attack the cancer and may interfere with the ability of tumor cells to grow and spread. Giving ipilimumab and nivolumab may lower the chance of recurrent glioblastoma with high number of mutations from growing or spreading compared to usual care (surgery or chemotherapy).

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine whether the combination of ipilimumab and nivolumab increases the tumor response rate assessed by modified Response Assessment in Neuro-Oncology (RANO) Criteria in patients with hypermutated recurrent glioblastoma.

SECONDARY OBJECTIVES:

I. Estimate the overall survival distribution, median survival, and one-year survival rate of patients with hypermutated, recurrent glioblastoma who are treated with ipilimumab and nivolumab.

II. Estimate the progression-free survival distribution and median progression-free survival of patients with hypermutated, recurrent glioblastoma who are treated with ipilimumab and nivolumab.

III. Determine the adverse event profile of patients with hypermutated, recurrent glioblastoma who are treated with ipilimumab and nivolumab.

EXPLORATORY OBJECTIVES:

I. Test whether PD-L1 or immunologic infiltrate in the tumor microenvironment are associated with objective tumor response, overall survival, progression-free survival, tumor mutational burden, or rates of grade 3 or higher adverse events.

II. Test whether MGMT status, microsatellite instability (MSI) status, mutational signatures, or amount of tumor mutational burden (TMB) including germline analysis are associated with objective tumor response, overall survival, progression-free survival, or rates of grade 3 or higher adverse events.

III. Evaluate associations between exome and transcriptome gene levels with objective tumor response, overall survival, progression-free survival, rates of grade 3 or higher adverse events.

IV. Evaluate associations between the gut microbiome and objective tumor response.

V. Response rate using immunotherapy (i)RANO.

OUTLINE:

Patients receive nivolumab intravenously (IV) over 30 minutes and ipilimumab IV over 30 minutes on day 1. Treatment repeats every 3 weeks for 4 cycles in the absence of disease progression or unacceptable toxicity. Patients then receive nivolumab IV over 30 minutes on day 1. Cycles repeat every 4 weeks in the absence of disease progression or unacceptable toxicity. Patients also undergo magnetic resonance imaging (MRI) throughout the study.

After completion of study treatment, patients without disease progression are followed every 8 weeks until disease progression, then every 3 months for up to 3 years. Patients with disease progression after completion of study treatment are followed every 3 months for up to 3 years.

ELIGIBILITY:
Inclusion Criteria:

* PRE-REGISTRATION ELIGIBILITY CRITERIA:
* Histologically confirmed glioblastoma (World Health Organization [WHO] grade IV) presenting at first or second recurrence including secondary glioblastoma

  * Glioblastoma IDH-wildtype central nervous system (CNS) WHO grade 4

    * Diffuse, astrocytic glioma IDH-wildtype with one or more of the following histological or genetic features: microvascular proliferation, necrosis, TERT promoter mutation, EGFR gene amplification, +7/-10 chromosome copy-number changes
  * Astrocytoma, IDH-mutant CNS WHO grade 4

    * Diffuse astrocytic glioma IDH-mutant (with frequent ATRX and/or TP53 mutation and absence of 1p/19q codeletion), with necrosis and/or microvascular proliferation or one with lower grade histological features displaying homozygous deletion of CDKN2A and/or CDKN2B
  * NOTE: The eligibility criteria were changed to include the new diagnostic language from the WHO 2021 pathology classification change. The above diagnoses therefore reflect the change and include the entities that were previously eligible but now carry updated pathologic classification
* Presence of measurable disease, as defined by a bidimensionally measurable lesion on magnetic resonance imaging (MRI) with a minimum diameter of 10 mm in both dimensions, prior to resection or biopsy of recurrent tumor
* Tissue available from surgical resection or biopsy of recurrent tumor =< 28 days prior to pre-registration, or planned surgery or biopsy of recurrent tumor =< 28 days after pre-registration
* Does not require > 4 mg dexamethasone beyond the perioperative period defined as the time =< 2 weeks after surgical procedure
* No active autoimmune disease or history of autoimmune disease

  * These include but are not limited to patients with a history of immune related neurologic disease, multiple sclerosis, autoimmune (demyelinating) neuropathy, Guillain-Barre syndrome, myasthenia gravis; systemic autoimmune disease such as systemic lupus erythematosus (SLE), connective tissue diseases, scleroderma, inflammatory bowel disease (IBD), Crohn's, ulcerative colitis, hepatitis; and patients with a history of toxic epidermal necrolysis (TEN), Stevens-Johnson syndrome, or phospholipid syndrome should be excluded because of the risk of recurrence or exacerbation of disease
  * Patients with vitiligo, endocrine deficiencies including thyroiditis managed with replacement hormones including physiologic corticosteroids are eligible. Patients with rheumatoid arthritis and other arthropathies, Sjogren's syndrome and psoriasis controlled with topical medication and patients with positive serology, such as antinuclear antibodies (ANA), anti-thyroid antibodies should be evaluated for the presence of target organ involvement and potential need for systemic treatment but should otherwise be eligible
* No prior treatment with checkpoint blockade therapies (anti-CTLA4, anti-PD1/PD-L1) or bevacizumab
* No prior treatment with laser ablation at the time of recurrent tumor tissue sampling. Patients who have previously undergone laser ablation >= 4 months prior to recurrent tumor tissue sampling can be included
* Age >= 18 years
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2
* Able to undergo brain MRI with contrast
* Absolute neutrophil count >= 1500/mm^3
* Platelet count >= 100,000/mm^3
* Total bilirubin =< 1.5 x upper limit of normal (ULN)

  * If Gilbert syndrome, then total bilirubin =< 3 x ULN
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) =< 2.0 x ULN
* Creatinine =< 1.5 x ULN OR creatinine clearance (CrCl) >= 50 mL/min (if using the Cockcroft-Gault formula)
* History of active malignancy (outside of the patient's glioblastoma) that has required treatment within the previous 2 years. Participant with prior history of in situ cancer or basal or squamous cell skin cancer are eligible
* REGISTRATION ELIGIBILITY CRITERIA: Tissue obtained from biopsy or resection at first or second recurrence exhibits TMB >= 10 on FoundationOne CDx testing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Estimated)
Dates: Start 2020-12-24 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Overall response rate | Up to 32 months
  Assessed by the Response Assessment in Neuro-Oncology Criteria (RANO). The proportion of patients who have a confirmed tumor response will be computed as the number of patients with a confirmed complete response or confirmed partial response as determined by RANO criteria divided by the number of evaluable patients, which are eligible patients who have measurable disease and completed one cycle of treatment. Will be estimated with a binomial point estimate that will be computed as the number of responses divided by the number of evaluable patients. Exact 95% binomial confidence intervals will be generated and reported.

SECONDARY OUTCOMES:
Overall survival (OS) | From the time of treatment initiation until death from any cause, assessed up to 3 years
  Will be summarized using Kaplan-Meier (KM) estimators. Survival curves will be generated from the KM estimators. KM estimates will be determined for the median OS as well as the 12-month OS rates. Confidence intervals will be provided for the median values as well as the one-year rates.
Progression-free survival (PFS) | From the time of treatment initiation until disease progression as measured using RANO criteria or death, whichever occurs first, assessed up to 3 years
  Will be summarized using KM estimators. Survival curves will be generated from the KM estimators. KM estimates will be determined for the median PFS as well as the 12-month PFS rates. Confidence intervals will be provided for the median values as well as the one-year rates.
Incidence of adverse events (AEs) | Up to 3 years
  The AEs will be summarized by the frequency and relative frequency of the maximum grade experienced by the patients for all recorded AEs. Adverse event data will be summarized by each observed AE with the number of patients who reported the AE as well as the proportion of patients with the AE.

CONTACTS AND LOCATIONS:
Overall Officials: Gavin P Dunn, Principal Investigator — Alliance for Clinical Trials in Oncology
Locations (416):
- United States (415):
  - Anchorage Associates in Radiation Medicine, Anchorage, Alaska
  - Anchorage Radiation Therapy Center, Anchorage, Alaska
  - Alaska Breast Care and Surgery LLC, Anchorage, Alaska
  - Alaska Oncology and Hematology LLC, Anchorage, Alaska
  - Alaska Women's Cancer Care, Anchorage, Alaska
  - Anchorage Oncology Centre, Anchorage, Alaska
  - Katmai Oncology Group, Anchorage, Alaska
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Cancer Center at Saint Joseph's, Phoenix, Arizona
  - Mayo Clinic Hospital in Arizona, Phoenix, Arizona
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mercy Hospital Fort Smith, Fort Smith, Arkansas
  - CHI Saint Vincent Cancer Center Hot Springs, Hot Springs, Arkansas
  - Mission Hope Medical Oncology - Arroyo Grande, Arroyo Grande, California
  - Providence Saint Joseph Medical Center/Disney Family Cancer Center, Burbank, California
  - Mercy Cancer Center - Carmichael, Carmichael, California
  - Mercy San Juan Medical Center, Carmichael, California
  - Mercy Cancer Center - Elk Grove, Elk Grove, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Mercy Cancer Center - Rocklin, Rocklin, California
  - Mercy Cancer Center - Sacramento, Sacramento, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Pacific Central Coast Health Center-San Luis Obispo, San Luis Obispo, California
  - Mission Hope Medical Oncology - Santa Maria, Santa Maria, California
  - Torrance Memorial Physician Network - Cancer Care, Torrance, California
  - Torrance Memorial Medical Center, Torrance, California
  - Woodland Memorial Hospital, Woodland, California
  - UCHealth University of Colorado Hospital, Aurora, Colorado
  - Rocky Mountain Cancer Centers-Boulder, Boulder, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - Rocky Mountain Cancer Centers-Penrose, Colorado Springs, Colorado
  - AdventHealth Porter, Denver, Colorado
  - CommonSpirit Cancer Center Mercy, Durango, Colorado
  - Mercy Medical Center, Durango, Colorado
  - Saint Anthony Hospital, Lakewood, Colorado
  - AdventHealth Littleton, Littleton, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - Rocky Mountain Cancer Centers-Longmont, Longmont, Colorado
  - AdventHealth Parker, Parker, Colorado
  - Saint Mary Corwin Medical Center, Pueblo, Colorado
  - Beebe Medical Center, Lewes, Delaware
  - Beebe South Coastal Health Campus, Millville, Delaware
  - Delaware Clinical and Laboratory Physicians PA, Newark, Delaware
  - Helen F Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Beebe Health Campus, Rehoboth Beach, Delaware
  - TidalHealth Nanticoke / Allen Cancer Center, Seaford, Delaware
  - Christiana Care Health System-Wilmington Hospital, Wilmington, Delaware
  - Holy Cross Hospital, Fort Lauderdale, Florida
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Low Country Cancer Care, Savannah, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Saint Alphonsus Cancer Care Center-Caldwell, Caldwell, Idaho
  - Kootenai Health - Coeur d'Alene, Coeur d'Alene, Idaho
  - Walter Knox Memorial Hospital, Emmett, Idaho
  - Saint Luke's Cancer Institute - Fruitland, Fruitland, Idaho
  - Idaho Urologic Institute-Meridian, Meridian, Idaho
  - Saint Luke's Cancer Institute - Meridian, Meridian, Idaho
  - Saint Alphonsus Cancer Care Center-Nampa, Nampa, Idaho
  - Saint Luke's Cancer Institute - Nampa, Nampa, Idaho
  - Kootenai Clinic Cancer Services - Post Falls, Post Falls, Idaho
  - Kootenai Clinic Cancer Services - Sandpoint, Sandpoint, Idaho
  - Saint Luke's Cancer Institute - Twin Falls, Twin Falls, Idaho
  - OSF Saint Anthony's Health Center, Alton, Illinois
  - Rush-Copley Medical Center, Aurora, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Memorial Hospital of Carbondale, Carbondale, Illinois
  - SIH Cancer Institute, Carterville, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - University of Illinois, Chicago, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Illinois CancerCare-Dixon, Dixon, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - NorthShore University HealthSystem-Evanston Hospital, Evanston, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Western Illinois Cancer Treatment Center, Galesburg, Illinois
  - NorthShore University HealthSystem-Glenbrook Hospital, Glenview, Illinois
  - NorthShore University HealthSystem-Highland Park Hospital, Highland Park, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - SSM Health Good Samaritan, Mount Vernon, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - OSF Saint Francis Radiation Oncology at Pekin, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - OSF Saint Francis Radiation Oncology at Peoria Cancer Center, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Valley Radiation Oncology, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - North Shore Medical Center, Skokie, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Springfield Memorial Hospital, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - The Carle Foundation Hospital, Urbana, Illinois
  - Illinois CancerCare - Washington, Washington, Illinois
  - Rush-Copley Healthcare Center, Yorkville, Illinois
  - Baptist Health Floyd, New Albany, Indiana
  - Mary Greeley Medical Center, Ames, Iowa
  - McFarland Clinic - Ames, Ames, Iowa
  - McFarland Clinic - Boone, Boone, Iowa
  - Saint Anthony Regional Hospital, Carroll, Iowa
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - UI Health Care Mission Cancer and Blood - West Des Moines Clinic, Clive, Iowa
  - Alegent Health Mercy Hospital, Council Bluffs, Iowa
  - Heartland Oncology and Hematology LLP, Council Bluffs, Iowa
  - Methodist Jennie Edmundson Hospital, Council Bluffs, Iowa
  - Greater Regional Medical Center, Creston, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Des Moines Clinic, Des Moines, Iowa
  - Broadlawns Medical Center, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Laurel Clinic, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - McFarland Clinic - Trinity Cancer Center, Fort Dodge, Iowa
  - UI Healthcare Mission Cancer and Blood - Fort Dodge, Fort Dodge, Iowa
  - McFarland Clinic - Jefferson, Jefferson, Iowa
  - McFarland Clinic - Marshalltown, Marshalltown, Iowa
  - Methodist West Hospital, West Des Moines, Iowa
  - Mercy Medical Center-West Lakes, West Des Moines, Iowa
  - Cancer Center of Kansas - Chanute, Chanute, Kansas
  - Cancer Center of Kansas - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas - El Dorado, El Dorado, Kansas
  - Central Care Cancer Center - Garden City, Garden City, Kansas
  - Central Care Cancer Center - Great Bend, Great Bend, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Cancer Center of Kansas-Kingman, Kingman, Kansas
  - Cancer Center of Kansas-Liberal, Liberal, Kansas
  - Cancer Center of Kansas-Manhattan, Manhattan, Kansas
  - Cancer Center of Kansas - McPherson, McPherson, Kansas
  - Cancer Center of Kansas - Newton, Newton, Kansas
  - Cancer Center of Kansas - Parsons, Parsons, Kansas
  - Cancer Center of Kansas - Pratt, Pratt, Kansas
  - Cancer Center of Kansas - Salina, Salina, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Ascension Via Christi Hospitals Wichita, Wichita, Kansas
  - Cancer Center of Kansas - Wichita, Wichita, Kansas
  - Cancer Center of Kansas - Winfield, Winfield, Kansas
  - Flaget Memorial Hospital, Bardstown, Kentucky
  - Commonwealth Cancer Center-Corbin, Corbin, Kentucky
  - Baptist Health Lexington, Lexington, Kentucky
  - Saint Joseph Radiation Oncology Resource Center, Lexington, Kentucky
  - Saint Joseph Hospital East, Lexington, Kentucky
  - Saint Joseph London, London, Kentucky
  - Jewish Hospital, Louisville, Kentucky
  - Baptist Health Louisville, Louisville, Kentucky
  - Saints Mary and Elizabeth Hospital, Louisville, Kentucky
  - UofL Health Medical Center Northeast, Louisville, Kentucky
  - Jewish Hospital Medical Center South, Shepherdsville, Kentucky
  - Ochsner LSU Health Monroe Medical Center, Monroe, Louisiana
  - LSU Health Sciences Center at Shreveport, Shreveport, Louisiana
  - Trinity Health Saint Joseph Mercy Hospital Ann Arbor, Ann Arbor, Michigan
  - Bronson Battle Creek, Battle Creek, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Brighton, Brighton, Michigan
  - Trinity Health Medical Center - Brighton, Brighton, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Canton, Canton, Michigan
  - Trinity Health Medical Center - Canton, Canton, Michigan
  - Caro Cancer Center, Caro, Michigan
  - Chelsea Hospital, Chelsea, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Chelsea Hospital, Chelsea, Michigan
  - Hematology Oncology Consultants-Clarkston, Clarkston, Michigan
  - Newland Medical Associates-Clarkston, Clarkston, Michigan
  - Henry Ford Health Saint John Hospital, Detroit, Michigan
  - Henry Ford River District Hospital, East China Township, Michigan
  - Cancer Hematology Centers - Flint, Flint, Michigan
  - Genesee Hematology Oncology PC, Flint, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Corewell Health Grand Rapids Hospitals - Butterworth Hospital, Grand Rapids, Michigan
  - Corewell Health Grand Rapids Hospitals - Helen DeVos Children's Hospital, Grand Rapids, Michigan
  - Trinity Health Grand Rapids Hospital, Grand Rapids, Michigan
  - Henry Ford Saint John Hospital - Academic, Grosse Pointe Woods, Michigan
  - Henry Ford Saint John Hospital - Breast, Grosse Pointe Woods, Michigan
  - Henry Ford Saint John Hospital - Van Elslander, Grosse Pointe Woods, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Beacon Kalamazoo Cancer Center, Kalamazoo, Michigan
  - Beacon Kalamazoo, Kalamazoo, Michigan
  - University of Michigan Health - Sparrow Lansing, Lansing, Michigan
  - Hope Cancer Clinic, Livonia, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - Henry Ford Saint John Hospital - Macomb Medical, Macomb, Michigan
  - Henry Ford Warren Hospital - Breast Macomb, Macomb, Michigan
  - Saint Mary's Oncology/Hematology Associates of Marlette, Marlette, Michigan
  - Trinity Health Muskegon Hospital, Muskegon, Michigan
  - Corewell Health Lakeland Hospitals - Niles Hospital, Niles, Michigan
  - Cancer and Hematology Centers of Western Michigan - Norton Shores, Norton Shores, Michigan
  - Hope Cancer Center, Pontiac, Michigan
  - Michigan Healthcare Professionals Pontiac, Pontiac, Michigan
  - Newland Medical Associates-Pontiac, Pontiac, Michigan
  - Trinity Health Saint Joseph Mercy Oakland Hospital, Pontiac, Michigan
  - Corewell Health Reed City Hospital, Reed City, Michigan
  - Henry Ford Rochester Hospital, Rochester Hills, Michigan
  - Corewell Health William Beaumont University Hospital, Royal Oak, Michigan
  - MyMichigan Medical Center Saginaw, Saginaw, Michigan
  - Oncology Hematology Associates of Saginaw Valley PC, Saginaw, Michigan
  - Corewell Health Lakeland Hospitals - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Corewell Health Lakeland Hospitals - Saint Joseph Hospital, Saint Joseph, Michigan
  - Bhadresh Nayak MD PC-Sterling Heights, Sterling Heights, Michigan
  - MyMichigan Medical Center Tawas, Tawas City, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Corewell Health Beaumont Troy Hospital, Troy, Michigan
  - Advanced Breast Care Center PLLC, Warren, Michigan
  - Henry Ford Health Warren Hospital, Warren, Michigan
  - Henry Ford Madison Heights Hospital - Breast, Warren, Michigan
  - Henry Ford Warren Hospital - GLCMS, Warren, Michigan
  - Macomb Hematology Oncology PC, Warren, Michigan
  - Saint Mary's Oncology/Hematology Associates of West Branch, West Branch, Michigan
  - University of Michigan Health - West, Wyoming, Michigan
  - Huron Gastroenterology PC, Ypsilanti, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology Ann Arbor Campus, Ypsilanti, Michigan
  - Sanford Joe Lueken Cancer Center, Bemidji, Minnesota
  - Essentia Health Saint Joseph's Medical Center, Brainerd, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Minnesota Oncology - Burnsville, Burnsville, Minnesota
  - Cambridge Medical Center, Cambridge, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Essentia Health - Deer River Clinic, Deer River, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Essentia Health Hibbing Clinic, Hibbing, Minnesota
  - Fairview Clinics and Surgery Center Maple Grove, Maple Grove, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Health Partners Inc, Minneapolis, Minnesota
  - Monticello Cancer Center, Monticello, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - Fairview Northland Medical Center, Princeton, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Coborn Cancer Center at Saint Cloud Hospital, Saint Cloud, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Essentia Health Sandstone, Sandstone, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Sanford Thief River Falls Medical Center, Thief River Falls, Minnesota
  - Essentia Health Virginia Clinic, Virginia, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Sanford Cancer Center Worthington, Worthington, Minnesota
  - Fairview Lakes Medical Center, Wyoming, Minnesota
  - Mercy Oncology and Hematology - Clayton-Clarkson, Ballwin, Missouri
  - Central Care Cancer Center - Bolivar, Bolivar, Missouri
  - Mercy Cancer Center - Cape Girardeau, Cape Girardeau, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - Parkland Health Center - Farmington, Farmington, Missouri
  - MU Health Care Goldschmidt Cancer Center, Jefferson City, Missouri
  - Freeman Health System, Joplin, Missouri
  - Mercy Hospital Joplin, Joplin, Missouri
  - Mercy Clinic-Rolla-Cancer and Hematology, Rolla, Missouri
  - Phelps Health Delbert Day Cancer Institute, Rolla, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Mercy Infusion Center - Chippewa, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital South, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - BJC Outpatient Center at Sunset Hills, Sunset Hills, Missouri
  - Mercy Hospital Washington, Washington, Missouri
  - Community Hospital of Anaconda, Anaconda, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Bozeman Health Deaconess Hospital, Bozeman, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Logan Health Medical Center, Kalispell, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - Community Medical Center, Missoula, Montana
  - Nebraska Cancer Specialists/Oncology Hematology West PC, Grand Island, Nebraska
  - CHI Health Good Samaritan, Kearney, Nebraska
  - Saint Elizabeth Regional Medical Center, Lincoln, Nebraska
  - Cancer Partners of Nebraska, Lincoln, Nebraska
  - Nebraska Cancer Specialists/Oncology Hematology West PC - MECC, Omaha, Nebraska
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Oncology Associates PC, Omaha, Nebraska
  - Alegent Health Immanuel Medical Center, Omaha, Nebraska
  - Alegent Health Bergan Mercy Medical Center, Omaha, Nebraska
  - Alegent Health Lakeside Hospital, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - Midlands Community Hospital, Papillion, Nebraska
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - Morristown Medical Center, Morristown, New Jersey
  - Jersey Shore Medical Center, Neptune City, New Jersey
  - Capital Health Medical Center-Hopewell, Pennington, New Jersey
  - Overlook Hospital, Summit, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - Randolph Hospital, Asheboro, North Carolina
  - Messino Cancer Centers, Asheville, North Carolina
  - Cone Health Cancer Center at Alamance Regional, Burlington, North Carolina
  - Cone Health Cancer Center, Greensboro, North Carolina
  - Cone Health Cancer Center at Drawbridge Parkway, Greensboro, North Carolina
  - ECU Health Medical Center, Greenville, North Carolina
  - Cone Heath Cancer Center at Mebane, Mebane, North Carolina
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Essentia Health Cancer Center-South University Clinic, Fargo, North Dakota
  - Sanford South University Medical Center, Fargo, North Dakota
  - Southpointe-Sanford Medical Center Fargo, Fargo, North Dakota
  - Sanford Medical Center Fargo, Fargo, North Dakota
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - Miami Valley Hospital South, Centerville, Ohio
  - University of Cincinnati Cancer Center-UC Medical Center, Cincinnati, Ohio
  - Good Samaritan Hospital - Cincinnati, Cincinnati, Ohio
  - Bethesda North Hospital, Cincinnati, Ohio
  - TriHealth Cancer Institute-Westside, Cincinnati, Ohio
  - TriHealth Cancer Institute-Anderson, Cincinnati, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Premier Blood and Cancer Center, Dayton, Ohio
  - Dayton Physician LLC - Englewood, Dayton, Ohio
  - Miami Valley Hospital North, Dayton, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Miami Valley Cancer Care and Infusion, Greenville, Ohio
  - Greater Dayton Cancer Center, Kettering, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - University of Cincinnati Cancer Center-West Chester, West Chester, Ohio
  - Cancer Centers of Southwest Oklahoma Research, Lawton, Oklahoma
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Mercy Hospital Oklahoma City, Oklahoma City, Oklahoma
  - Saint Alphonsus Cancer Care Center-Baker City, Baker City, Oregon
  - Saint Charles Health System, Bend, Oregon
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Providence Cancer Institute Clackamas Clinic, Clackamas, Oregon
  - Bay Area Hospital, Coos Bay, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Saint Alphonsus Cancer Care Center-Ontario, Ontario, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Saint Charles Health System-Redmond, Redmond, Oregon
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - Christiana Care Health System-Concord Health Center, Chadds Ford, Pennsylvania
  - Pocono Medical Center, East Stroudsburg, Pennsylvania
  - Lehigh Valley Hospital-Hazleton, Hazleton, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - Reading Hospital, West Reading, Pennsylvania
  - Gibbs Cancer Center-Pelham, Greer, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Saint Joseph Regional Cancer Center, Bryan, Texas
  - Parkland Memorial Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - Inova Schar Cancer Institute, Fairfax, Virginia
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Providence Regional Cancer System-Aberdeen, Aberdeen, Washington
  - PeaceHealth Saint Joseph Medical Center, Bellingham, Washington
  - Highline Medical Center-Main Campus, Burien, Washington
  - Providence Regional Cancer System-Centralia, Centralia, Washington
  - Swedish Cancer Institute-Edmonds, Edmonds, Washington
  - Saint Elizabeth Hospital, Enumclaw, Washington
  - Providence Regional Cancer Partnership, Everett, Washington
  - Saint Francis Hospital, Federal Way, Washington
  - Swedish Cancer Institute-Issaquah, Issaquah, Washington
  - Kadlec Clinic Hematology and Oncology, Kennewick, Washington
  - Providence Regional Cancer System-Lacey, Lacey, Washington
  - Saint Clare Hospital, Lakewood, Washington
  - PeaceHealth Saint John Medical Center, Longview, Washington
  - Jefferson Healthcare, Port Townsend, Washington
  - Harrison HealthPartners Hematology and Oncology-Poulsbo, Poulsbo, Washington
  - Pacific Gynecology Specialists, Seattle, Washington
  - Swedish Medical Center-Ballard Campus, Seattle, Washington
  - Swedish Medical Center-Cherry Hill, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - PeaceHealth United General Medical Center, Sedro-Woolley, Washington
  - Providence Regional Cancer System-Shelton, Shelton, Washington
  - Saint Michael Cancer Center, Silverdale, Washington
  - Franciscan Research Center-Northwest Medical Plaza, Tacoma, Washington
  - Northwest Medical Specialties PLLC, Tacoma, Washington
  - PeaceHealth Southwest Medical Center, Vancouver, Washington
  - Providence Saint Mary Regional Cancer Center, Walla Walla, Washington
  - Providence Regional Cancer System-Yelm, Yelm, Washington
  - United Hospital Center, Bridgeport, West Virginia
  - WVUH-Berkely Medical Center, Martinsburg, West Virginia
  - West Virginia University Healthcare, Morgantown, West Virginia
  - Camden Clark Medical Center, Parkersburg, West Virginia
  - Duluth Clinic Ashland, Ashland, Wisconsin
  - Mayo Clinic Health System-Eau Claire Clinic, Eau Claire, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - ProHealth D N Greenwald Center, Mukwonago, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - ProHealth Oconomowoc Memorial Hospital, Oconomowoc, Wisconsin
  - ProHealth Waukesha Memorial Hospital, Waukesha, Wisconsin
  - UW Cancer Center at ProHealth Care, Waukesha, Wisconsin
  - Billings Clinic-Cody, Cody, Wyoming
  - Welch Cancer Center, Sheridan, Wyoming
- Pan American Center for Oncology Trials LLC, San Juan, Puerto Rico

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page
URL: https://grants.nih.gov/policy/sharing.htm